CLINICAL TRIAL: NCT06839391
Title: Effect of Hyaluronidase in Different Doses Added to Bupivacaine on TAB Block Quality During CS
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Mohamed said MOSTAFA elmeligy, anesthesia lecturer, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TAB BLOCK QAULITY
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Tab Block Qaulity
Keywords: hyaluronidase-bupivacaine-TAB block
MeSH Terms: interventions — Hyaluronoglucosaminidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group I (Experimental): After skin closure, they got TAB block with 20 cc of 0.25 percent bupivacaine on each side without any adjuvant.
  Interventions: Drug: Hyaluronidase
- group II (Experimental): obtained After the skin was closed, we received TAB block with 20 ml of 0.25% bupivacaine and 5 ml of 0.9% normal saline containing 500 IU (100 IU/ml) of hyaluronidase (Hynidase) as an adjuvant on each side.
  Interventions: Drug: Hyaluronidase
- GROUP III (Experimental): obtained After the skin was closed, we received TAB block with 20 ml of 0.25% bupivacaine and 5 ml of 0.9% normal saline containing 1000 IU (200 IU/ml) hyaluronidase (Hynidase) as an adjuvant on each side.
  Interventions: Drug: Hyaluronidase

INTERVENTIONS:
Drug: Hyaluronidase — Effect of hyaluronidases in different doses added to bupivacaine on quality of ultrasound-guided TAB block during CS ,

SUMMARY:
evaluate the efficacy of hyaluronidase in different doses as an adjuvant to bupivacaine in ultrasound-guided TAB block during CS

DETAILED DESCRIPTION:
Hyaluronidase acts by catalyzing the hydrolysis of hyaluronan, decreased its viscosity, and enchasing the tissue permeability. So, this makes it a suitable additive for other drugs to speed up their distribution and delivery especially in ophthalmic surgery. Several studies showed that multiple injection techniques of TAB block were more successful with a faster onset of anesthesia and higher success rates, with a change in the incidence of complications.

This double-blinded randomized prospective study was conducted to evaluate the efficacy of hyaluronidase in different doses as an adjuvant to bupivacaine in ultrasound-guided TAB block during CS . The primary outcome of this study was the duration of sensory block, while secondary outcomes included the onset of sensory block, success rate, total doses of intraoperative rescue analgesia, number of patients needed for postoperative rescue analgesia, and complications.

ELIGIBILITY:
Inclusion Criteria:

* pregnant 20-45 y medical free

Exclusion Criteria:

* • Hepatic.

  * Renal.
  * Diabetic.
  * Hypertensive.
  * Cardiovascular dysfunction.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale | 2-6-10-16-24 hours postoperatively
  postoperatively pain assesment

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Keeler JF, Simpson KH, Ellis FR, Kay SP. Effect of addition of hyaluronidase to bupivacaine during axillary brachial plexus block. Br J Anaesth. 1992 Jan;68(1):68-71. doi: 10.1093/bja/68.1.68. PMID 1739571
- [Background] Koh WU, Min HG, Park HS, Karm MH, Lee KK, Yang HS, Ro YJ. Use of hyaluronidase as an adjuvant to ropivacaine to reduce axillary brachial plexus block onset time: a prospective, randomised controlled study. Anaesthesia. 2015 Mar;70(3):282-9. doi: 10.1111/anae.12879. Epub 2014 Oct 28. PMID 25347936
- [Background] Kumar CM, Macachor J. Hyaluronidase for brachial plexus block. Anaesthesia. 2015 Sep;70(9):1097-8. doi: 10.1111/anae.13186. No abstract available. PMID 26263864